CLINICAL TRIAL: NCT03674658
Title: An Open-Label Randomized Study of Propafenone in the Treatment of Atrial Fibrillation
Brief Title: Propafenone in the Treatment of Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TSH Biopharm Corporation Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TSHRH1801-P
Record Dates: First submitted 2018-09-14; First posted 2018-09-17 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Propafenone

STUDY DESIGN:
Intervention Model Description: Group A: Rhynorm (A drug) Group B: Rytmonorm (B drug)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A drug (Experimental): Rhynorm(A drug)
  Interventions: Drug: Propafenone
- B drug (Active Comparator): Rytmonorm (B drug)
  Interventions: Drug: Propafenone

INTERVENTIONS:
Drug: Propafenone — oral, TID
  Other Names: A drug: Rhynorm; B drug: Rytmonorm

SUMMARY:
This is a open label randomized, multi-center study conducted in Taiwan. The study aims to evaluate the effectiveness and safety of oral Rhynorm (A drug) and Rytmonorm (B drug) for the conversion of paroxysmal AF and is designed to evaluate the improvement in sinus rhythm restoration after the treatment with Rhynorm (A drug) and Rytmonorm (B drug) for 24 weeks.

DETAILED DESCRIPTION:
This is a open label randomized, multi-center study conducted in Taiwan. The study aims to evaluate the effectiveness and safety of oral Rhynorm (A drug) and Rytmonorm (B drug) for the conversion of paroxysmal AF and is designed to evaluate the improvement in sinus rhythm restoration after the treatment with Rhynorm (A drug) and Rytmonorm (B drug) for 24 weeks.

This study comprised of three phases: a screening phase, a washout run-in qualifying phase lasting about 7 days, and a treatment phase of 24 weeks. A total of 60 evaluable subjects is planned to be enrolled. With an estimation of 20% dropout rate, 72 patients will be enrolled to reach 60 evaluable patients at the end of study. After screening for eligibility, the eligible subjects will be randomly assigned to either of the two gruop. The two-group are shown in the following table.

Group Treatment Drug Group A Rhynorm (A drug) Group B Rytmonorm (B drug) Patients with arrhythmia will be screened for eligibility after providing informed consent. Patients present with the symptoms of arrhythmia after withdrawn from other prohibited anti-AF agents for at least 7 days and completed run-in period event recorded will be qualified for entering this study and will be randomized to Rhynorm (A drug) treatment group or Rytmonorm (B drug) reference drud group in a 1:1 ratio.

The clinical evaluation will be recorded during the study period. Before treating with Rhynorm (A drug) and Rytmonorm (B drug), the physical examination and condition will be tracked and recorded for at least 7 days as the historical data.

During the treatment period, the subjects still had a routine OPD visit. Record symptom event and event recorder monitoring on OPD visit.

Safety assessments on all randomized subjects include adverse events, vital signs, and laboratory tests (hematology and biochemistry). Any adverse events, symptom events and concomitant medications/therapies will be recorded on the CRFs throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are 20~80 years of age
2. Recurrent AF patients
3. Patients with paroxysmal atrial fibrillation
4. Patients diagnosed with one of the ECG monitoring within 12 months prior screening visit:

   1. 12-lead electrocardiogram
   2. ECG used to make a 30 second one of recording
   3. 24 hours ECG (Holter Monitor)
   4. Long term ECG (Event Monitor)
5. Patient may be receiving stable dose of propafenone since at least 4 weeks prior screening visit.
6. Agree to and are able to follow the study procedures
7. Understand the nature of the study, and have signed informed consent forms

Exclusion Criteria:

1. Permanent or persistent AF
2. Any of the following heart disease:

   1. New York Heart Association class III or IV angina pectoris or heart failure
   2. previous electrocardiographic evidence of second- or third-degree atrioventricular block;
   3. Sinus node disease, AV conduction disturbance or bundle branch block in the absence of an artificial pacemaker
   4. Hemodynamic moderate valvular heart disease (stenosis and/or incompetent; regurgitation)
   5. Brugada syndrome
   6. Left ventricular EF< 50%
   7. Acute myocardial infarction or unstable angina within the previous 12 months
   8. Cardiogenic shock (excluding arrhythrmia shock) within the previous 12 months
   9. Acute pericarditis or myocarditis within the previous 6 months
   10. Cardiac or thoracic surgery within the previous 6 months
3. Symptomatic Bradycardia (heart rate less than 50 beats per minute)
4. Hemodynamic instability, defined as hypotension (SBP < 90 mm Hg)
5. Hyperthyroidism
6. Bronchospastic disorders or severe obstructive pulmonary disease
7. Correctable AF for other reasons
8. Marked electrolyte imbalance
9. Patients with clinically significant abnormalities in the following laboratory parameters:

   1. AST or ALT ≥ 3X upper limit of normal (ULN)
   2. Total bilirubin ≥ 2X ULN
   3. Creatinine ≥ 2.5 mg/dL
   4. Hemoglobin < 10 g/dL
   5. Platelet < 100,000/uL
10. Patients with known contraindication or history of allergy to Propafenone.
11. Female patients who are pregnant or lactating.
12. Female patients of child-bearing potentiality who do not agree to use an effective method of contraception during the study
13. Patients currently participating in any drug related clinical trial within 30 days
14. Patients with propagating factor (e.g. Alcohol Abuse induced AF)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2019-07-11 (Actual); Primary Completion 2021-08-17 (Actual); Study Completion 2021-08-17 (Actual)

PRIMARY OUTCOMES:
proportion of patients with recurrent AF | 24 weeks treatment
  To compare the effect of Rhynorm (A drug) and Rytmonorm (B drug) over 24 weeks of treatment based on the proportion of patients with recurrent AF

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chin CG, Hsieh YC, Lin WS, Lin YJ, Chiou CW, Lin TH, Huang CL, Hung Y, Lin YK, Chang SL, Yeh TC, Lee HC, Lai WT, Hsieh MH. An open-label randomized noninferior study of generic name and brand name of propafenone for rhythm control in patients with paroxysmal atrial fibrillation. J Chin Med Assoc. 2023 May 1;86(5):472-478. doi: 10.1097/JCMA.0000000000000903. Epub 2023 Feb 17. PMID 36800262